CLINICAL TRIAL: NCT05655091
Title: Can Continuous Infusion Coupled With Therapeutic Drug Monitoring Optimize Flucloxacillin and Cefazolin Target Attainment Compared to Standard Intermittent Bolus Dosing in Patients With Complicated Staphylococcus Aureus Infections? A Randomized, Controlled Interventional Pilot Trial.
Brief Title: Target Attainment of Continuous Infusion Flucloxacillin and Cefazolin Coupled With TDM vs. Standard of Care Treatment in Patients With Complicated S. Aureus Infection
Acronym: TARGET III
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01708; am21Osthoff
Record Dates: First submitted 2022-11-30; First posted 2022-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Complicated Staphylococcus Aureus (S. Aureus) Infections (CSAI)
Keywords: Therapeutic drug monitoring (TDM); Flucloxacillin (FLU); Cefazolin (CZO); β-lactam antibiotics; antibiotic plasma concentration; standard intermittent bolus administration; continuous infusion; Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections; Infections

STUDY DESIGN:
Intervention Model Description: Single-centre, randomised, controlled, interventional pilot trial
Masking Description: There will be no blinding in this study. The antibiotic concentrations in the control group will be measured but not communicated to the study team or the treating physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): Subjects randomized into the intervention group will receive FLU or CZO respectively as continuous infusion as soon as targeted S. aureus treatment is initiated (+24h). The choice of antibiotic is determined by the treating physician in accordance to the recommendations of the infectious diseases (ID) specialists. The loading dose and dose adjustments of FLU and CZO will be determined by the use of a pharmacokinetic modelling application. The maximum daily dose will not exceed the daily licensed dose according to the Summary of Product Characteristics (SmPC).
  Interventions: Drug: FLU or CZO as continuous infusion
- control group (Active Comparator): Subjects randomized to the control group will receive standard of care intermittent bolus infusion FLU or CZO dosed according to the recommendations of the ID specialist and treating physician. Drug concentration will be analysed directly, but the results will not be communicated to the study team or a physician involved in the treatment of the patient. No TDM-guided dose adjustment will be performed in the control group.
  Interventions: Drug: standard FLU or CZO intermittent bolus administration

INTERVENTIONS:
Drug: FLU or CZO as continuous infusion — Continuous infusion FLU or CZO coupled with real-time TDM and subsequent dose adjustment. A loading dose will be administered prior to the first continuous infusion. The loading dose (maximum of 2g as licensed according to the SmPC) and the dose of the continuous infusion will be calculated according to a pharmacokinetic model taking into account patient's characteristics (e.g. age, sex) and the measured drug concentration. The maximum daily dose of FLU and CZO will not exceed 12 grams per day according to the SmPC.
  Arms: intervention group
Drug: standard FLU or CZO intermittent bolus administration — Standard FLU or CZO intermittent bolus administration according to the local guidelines adjusted to the renal function without TDM-guided dose adjustment.
  Arms: control group

SUMMARY:
This prospective randomized, controlled interventional pilot trial, aims to compare the achievement of the optimal target concentration with continuously administered flucloxacillin (FLU) or cefazolin (CZO) coupled with TDM and subsequent dose adjustment versus standard of care (intermittent bolus application without TDM-guidance) in patients with complicated Staphylococcus aureus (S. aureus) infections (CSAI). The overall goal is to individualize and optimize antibiotic treatment in a very vulnerable group of patients overcoming the standard strategy of "one-dose-fits-all".

DETAILED DESCRIPTION:
Therapeutic drug monitoring (TDM) has recently been established as one of the cornerstones to individualize treatment of β-lactam antibiotics. It is particularly useful in patients hospitalized in the intensive care unit (ICU) being at risk to not achieve optimal antibiotic plasma concentrations due to a strongly altered metabolism. Along the same lines, continuous administration of β-lactam antibiotics instead of standard intermittent bolus administration may maintain drug concentrations in the target range throughout the dosing interval, and even contribute to a decrease in mortality. This prospective randomized, controlled interventional pilot trial, aims to compare the achievement of the optimal target concentration with continuously administered flucloxacillin (FLU) or cefazolin (CZO) coupled with TDM and subsequent dose adjustment versus standard of care (intermittent bolus application without TDM-guidance) in patients with complicated Staphylococcus aureus (S. aureus) infections (CSAI). The overall goal is to individualize and optimize antibiotic treatment in a very vulnerable group of patients overcoming the standard strategy of "one-dose-fits-all". The primary objective of this trial is to evaluate the achievement of the optimal pharmacological target concentration (100% fT 2 to 12 mg/L) in blood on day 3 after inclusion with continuous infusion FLU and CZO in combination with real-time TDM and subsequent dose adjustment, versus the current standard of care in patients with CSAI, and to estimate the effect size for future trials. To evaluate the PKPD of unbound FLU or CZO in the intervention versus the control group as measured by the following:

* Drug concentration at second or later TDM including the incidence of high (e.g. 100% fT>12 mg/L) and low concentrations (e.g. 100% fT<2mg/L)
* Incidence of potential drug-related toxicity during the course of treatment (e.g. nephrotoxicity, hepatotoxicity, neurotoxicity)
* Time to optimal target attainment and percentage of days with optimal target attainment in relation to total study drug treatment duration
* Intra-individual variability in FLU und CZO total and unbound plasma concentrations
* Factors associated with pharmacological target attainment (e.g. kidney function, protein, albumin, age, sex, weight, concomitant medication)

Sub-study I:

- Evaluation of the pharmacological profile of penicillin in patients in whom treatment was changed from FLU or CZO to penicillin due to a penicillin susceptible S. aureus strain.

Sub-study II:

- Assessment of patient satisfaction, rest-activity rhythms and sleep quality by actigraphy, sleep diaries and questionnaire in patients admitted to a general ward.

Patients will be randomized in two parallel groups stratified to the use of FLU or CZO in a 1:1 ratio to be treated either by continuous infusion plus TDM and dose adjustment or by standard intermittent bolus application.

Drug concentrations will be measured at day 1, 3, 5, 7, 10 and thereafter two times weekly until treatment period is completed (i.e. up to 6 weeks) or until discharge. After discharge, TDM will be performed 1x/week if the patient is treated in the outpatient parenteral antibiotic treatment (OPAT) program but without any dose adjustments. Dose adjustments of FLU and CZO in the intervention group will be performed according to a pharmacokinetic modelling application that is based on the data of our previous studies TARGET [2] and TARGET II (unpublished data). In the control group, blood samples will be drawn and analysed directly, but the results will not be communicated to the study team or a physician involved in the treatment of the patient. No TDM-guided dose adjustment will be performed in the control group

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature. For patients, who are not able to sign consent, a physician not involved in the current study has to confirm that patient's interest and rights are guaranteed during participation in the current study. Subsequently, informed consent will be obtained as soon as possible from the patient or his/her legally authorised representative.
* Age ≥ 18 years
* CSAI which is defined as (i) blood stream infection (BSI) with S. aureus or (ii) deep-seated infections caused by S. aureus (e.g. osteoarticular infections, deep-seated abscesses) without BSI.
* Intended or active (less than 24 hours) treatment with FLU or CZO

Exclusion Criteria:

* Patients on hemodialysis or eGFR<10 ml/min as these patients have a special pharmacokinetic
* Patients on Cytosorb® therapy
* Patients with liver cirrhosis CHILD B and C
* Patients who are very likely to stop treatment with FLU or CZO in the next 48 hours as per treating physician (because of treatment failure, switch to oral medication, palliative care, allergy etc.) or who are very likely to be discharged or transferred to another hospital in the next 48 hours as per treating physician.
* Polymicrobial infection except concomitant isolation of a likely contaminant (e.g. Staphylococcus epidermidis or Cutibacterium acnes). If an additional pathogen is identified after inclusion of the patient into the study, the patient will remain in the study.
* CSAI caused by methicillin-resistant S. aureus (MRSA)
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Any uncontrolled or significant concurrent illness that would put the patient at a greater risk or limit compliance with the study requirements at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that attain the (FLU or CZO) target concentration (100% fT 2 to 12 mg/L) in blood. | On day 3 after inclusion
  For the assessment of the primary endpoint (100% fT 2 to 12 mg/L), the plasma concentration of FLU or CZO will be measured at day 3 after inclusion of the patient.

SECONDARY OUTCOMES:
Proportion of patients attaining the target (FLU or CZO) concentration at second TDM | At day 1, 3, 5, 7, 10 and thereafter two times weekly until treatment period is completed (i.e. up to 6 weeks) or until discharge
  Change in plasma concentration of FLU and CZO will be measured
Incidence of high (e.g. 100% fT>12 mg/L) (FLU or CZO) concentrations | At day 1, 3, 5, 7, 10 and thereafter two times weekly until treatment period is completed (i.e. up to 6 weeks) or until discharge
  Incidence of high (e.g. 100% fT>12 mg/L) (FLU or CZO) concentrations
Incidence of low concentrations (e.g. 100% fT<2mg/L) (FLU or CZO) concentrations | At day 1, 3, 5, 7, 10 and thereafter two times weekly until treatment period is completed (i.e. up to 6 weeks) or until discharge
  Incidence of low concentrations (e.g. 100% fT<2mg/L) (FLU or CZO) concentrations
Incidence of potential drug-related toxicity during the course of treatment (e.g. nephrotoxicity, hepatotoxicity, neurotoxicity) | From Day 0 (enrolment) until discharge (up to 6 weeks)
  Incidence of potential drug-related toxicity during the course of treatment (e.g. nephrotoxicity, hepatotoxicity, neurotoxicity)
Percentage of days with optimal target attainment in relation to total study treatment duration | From Day 0 (enrolment) until discharge (up to 6 weeks)
  Percentage of days with optimal target attainment in relation to total study treatment duration
Intra-individual variability in FLU und CZO total and unbound plasma concentrations | At day 1, 3, 5, 7, 10 and thereafter two times weekly until treatment period is completed (i.e. up to 6 weeks) or until discharge
  Intra-individual variability in FLU und CZO measured by change in plasma concentrations (total and unbound)

OTHER OUTCOMES:
Change in drug concentration of penicillin (in patients in whom treatment was changed from FLU or CZO to penicillin (Outcome of sub-study I)) | From Day 1 after enrolment until treatment period is completed (i.e. up to 6 weeks)
  Change in drug concentration of penicillin (in patients in whom treatment was changed from FLU or CZO to penicillin (Outcome of sub-study I))
Rest-activity rhythms in patients admitted to a general ward (Outcome of sub-study II) | From Day 0 (enrolment) until until end of treatment (up to 6 weeks)
  Rest-activity rhythms will be assessed by actigraphy. The actigraph will be worn on the non-dominant wrist all the time during the hospital stay. If patients are discharged, actigraphy will be continued as long as antibiotic treatment will be maintained.
Change in Sequential Organ Failure Assessment (SOFA) score | From Day 0 (enrolment) until day 10
  The Sequential Organ Failure Assessment (SOFA) score numerically quantifies the number and severity of failed organs. The SOFA score is made of 6 variables, each representing an organ system. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure).
Time to first negative blood culture | From Day 0 (enrolment) until discharge (approx. 2 weeks)
  Time to first negative blood culture
Change in inflammation parameters (C-reactive protein) | From Day 0 (enrolment) until end of treatment (up to 6 weeks)
  Change in inflammation parameters (C-reactive protein)
Change in All-cause mortality rate at day 30 and day 90 | At day 30 and day 90 after enrolment
  Change in All-cause mortality rate
Quality of life using the EuroQol™ 5D-5L Questionnaire | At day 90 after enrolment
  EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. (Score 0 to 100: 100 means the best health you can imagine. 0 means the worst health you can imagine).
Serious adverse events | From Day 1 after enrolment until three month follow-up
  All serious adverse events will be assessed and documented by the investigators according to seriousness, intensity, causal relationship with study treatment, action taken with study treatment (e.g. withdrawal), specific treatment for serious adverse event and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osthoff, PD Dr. med., Principal Investigator — University Hospital Basel, Division of Internal Medicine
Locations (1):
- University Hospital Basel, Division of Internal Medicine, Basel, Switzerland